CLINICAL TRIAL: NCT06894316
Title: Diaphragmatic-Based Complementary Training in Basketball: The Science Behind Pre-Activation of Inspiratory Muscles - A Randomized Trial
Brief Title: Inspiratory Muscle Warm-up Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Burak Karaca (Other)
Collaborators: University of Gaziantep (Other)
Responsible Party: Sponsor-Investigator, Burak Karaca, MSc. Burak KARACA, University of Gaziantep
Organization: University of Gaziantep (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2023-2; Gaziantep University (Registry Identifier: Social and Human Sciences Ethics Committee)
Record Dates: First submitted 2025-03-12; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Inspiratory Muscle Strength
Keywords: respiratory; exercise; accuracy; basketball
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Inspiratory Muscle Pre Activation Group (IMpa) (Experimental): The Powerbreathe brand device was used to perform inspiratory muscle pre-activation. Two sets of 30 breaths were carried out at 40% of each participant's maximal inspiratory mouth pressure (MIP), with a one-minute rest in between. MIP was measured once at the first session, and that value determined 40% and 5% for IMpa and IMPpa, respectively, in later visits. Participants were seated, wearing a nose clip, instructed to exhale forcefully, then inhale forcefully against a closed airway for one to three seconds. Measurements were repeated until values within 5 cmH₂O of each other were obtained, recording the best result in cmH₂O.
  Interventions: Device: Inspiratory muscle warm-up training
- Inspiratory Muscle Placebo Pre Activation Group (IMPpa) (Placebo Comparator): The Powerbreathe brand inspiratory muscle warm-up device was employed to facilitate an exercise regimen comprising two sets of 30 breaths, performed at an intensity of 5% of the participants' maximal inspiratory mouth pressure (MIP), with a one-minute interval between sets. This minimal load was intended as a placebo-like condition for inspiratory muscle usage.
  Interventions: Device: Placebo inspiratory muscle warm-up training
- Control Group (No Intervention): No warm-up protocol was applied to the control group.
- General Warm-up Group (Experimental): The participants engaged in a 10-minute jogging activity, which was followed by a 10-minute stretching exercise. Subsequently, the general warm-up protocol was completed with shooting drills tailored to the specific requirements of basketball, without inducing fatigue.
  Interventions: Other: General Warm-up Protocol

INTERVENTIONS:
Device: Inspiratory muscle warm-up training — The Powerbreathe brand device was used to perform inspiratory muscle pre-activation. Two sets of 30 breaths were carried out at 40% of each participant's maximal inspiratory mouth pressure (MIP), with a one-minute rest in between. MIP was measured once at the first session, and that value determined 40% and 5% for IMpa and IMPpa, respectively, in later visits. Participants were seated, wearing a nose clip, instructed to exhale forcefully, then inhale forcefully against a closed airway for one to three seconds. Measurements were repeated until values within 5 cmH₂O of each other were obtained, recording the best result in cmH₂O.
  Arms: Inspiratory Muscle Pre Activation Group (IMpa)
Other: General Warm-up Protocol — The participants engaged in a 10-minute jogging activity, which was followed by a 10-minute stretching exercise. Subsequently, the general warm-up protocol was completed with shooting drills tailored to the specific requirements of basketball, without inducing fatigue.
  Arms: General Warm-up Group
Device: Placebo inspiratory muscle warm-up training — The Powerbreathe brand inspiratory muscle warm-up device was employed to facilitate an exercise regimen comprising two sets of 30 breaths, performed at an intensity of 5% of the participants' maximal inspiratory mouth pressure (MIP), with a one-minute interval between sets. This minimal load was intended as a placebo-like condition for inspiratory muscle usage.
  Arms: Inspiratory Muscle Placebo Pre Activation Group (IMPpa)

SUMMARY:
The capacity of athletes to demonstrate their abilities to the fullest extent is contingent upon their physical fitness. Oxygen delivery and utilization become crucial during athletic pursuits, as muscle oxygen demand increases with exercise. The mechanical functioning of the respiratory system is largely dependent on the capacity of the respiratory muscles. For these reasons, inspiratory muscle pre-activation, which positively affects the efficiency of pulmonary circulation, increases the functional capacity of the respiratory muscles, reduces fatigue in the respiratory muscles, and plays a critical role in exercise physiology and athlete performance.

It has been demonstrated that inspiratory muscle exercises elicit a range of effects on performance. Studies show reductions in blood lactate levels among short-distance runners, thereby facilitating a positive enhancement in the post-performance recovery process, improve respiratory functions and both aerobic and anaerobic capacity in basketball players, positively affect performance in Olympic swimmers, increase performance in professional rowers and cyclists, enhance aerobic exercise performance in wheelchair basketball players, affect exercise performance in tennis players, increase performance in professional football players and handball players, affect shooting performance in archers, positively affect shot-hit performance in ice hockey players, and increase shot and drag-flick hit performance in hockey players. Nevertheless, there is a paucity of data concerning the impact of inspiratory muscle pre-activation on basketball performance. Many of these studies focus on longer-term training adaptations rather than a single short session of pre-activation.

The fundamental techniques of basketball can be classified into four main categories: passing, shooting, dribbling, and rebounding. Of these, shooting and passing are skills that require a high degree of accuracy in order to be performed effectively within the context of the game. A review of the literature reveals that training the inspiratory muscles is an effective method for improving athletic skills that require accuracy, as it enhances the stabilization of core muscles. However, the exact mechanism by which a brief inspiratory muscle pre-activation session might benefit precision-based movements remains under discussion. Therefore, the aim of this study was to examine whether a diaphragmatic-based method to prepare inspiratory muscles could improve passing, dribbling, and shooting among basketball players. By evaluating its immediate impact on key basketball tasks, we aim to clarify the value of such exercises in routine training.

DETAILED DESCRIPTION:
Participants The study involved 10 healthy male participants, aged between 18 and 25 years (mean age: 21.1 ± 2.42 years), who were engaged in competitive basketball. In order to be included in the study, the basketball players had to be free of both chronic and acute upper respiratory tract infections, as well as any chest diseases. The study was conducted in accordance with the ethical standards of the Declaration of Helsinki (52nd World Medical Association General Assembly, Edinburgh, Scotland, October 2000) and was approved by the Gaziantep University Social and Human Sciences Ethics Committee (approval number: 2023-2). Prior to the commencement of the study, informed consent was obtained from all participants.

Experimental design The study was designed according to a randomised, placebo-controlled, crossover structure. Following the initial interview, participants underwent a series of skill tests on four occasions throughout the course of the study, in accordance with established pre-activity steps. In the initial session, the participants were provided with general information about the research project. In addition to the measurement of age, height, and weight, an orientation session was conducted. In the subsequent four visits (1st, 2nd, 3rd, and 4th visits), randomised trials were carried out, including a control trial (no inspiratory pre-activation), an inspiratory muscle pre-activation (IMpa) at 40% MIP, a placebo inspiratory muscle pre-activation (IMPpa) at 5% MIP, and a general warm-up (GW) specific to basketball. The intensity values (40% for IMpa and 5% for IMPpa) were selected based on prior research indicating that moderate loading can meaningfully engage inspiratory muscles, whereas near-minimal loading provides an effective placebo condition.Following the random selection of participants by means of a card-drawing method, the Johnson basketball skill test and the American Alliance For Health, Physical Education, Recreation And Dance (AAHPERD) speed shooting test were administered.

Procedures Inspiratory muscle pre-activation trial (IMpa) The Powerbreathe brand device was used to perform inspiratory muscle pre-activation. Two sets of 30 breaths were carried out at 40% of each participant's maximal inspiratory mouth pressure (MIP), with a one-minute rest in between. MIP was measured once at the first session, and that value determined 40% and 5% for IMpa and IMPpa, respectively, in later visits. Participants were seated, wearing a nose clip, instructed to exhale forcefully, then inhale forcefully against a closed airway for one to three seconds. Measurements were repeated until values within 5 cmH₂O of each other were obtained, recording the best result in cmH₂O.

Placebo inspiratory muscle pre-activation trial (IMPpa) The Powerbreathe brand inspiratory muscle warm-up device was employed to facilitate an exercise regimen comprising two sets of 30 breaths, performed at an intensity of 5% of the participants' maximal inspiratory mouth pressure (MIP), with a one-minute interval between sets. This minimal load was intended as a placebo-like condition for inspiratory muscle usage.

General warm-up protocol (GW) The participants engaged in a 10-minute jogging activity, which was followed by a 10-minute stretching exercise. Subsequently, the general warm-up protocol was completed with shooting drills tailored to the specific requirements of basketball, without inducing fatigue.

Data collection Johnson basketball skill test In order to assess shooting ability, each participant was required to attempt to make as many successful shots as possible within a 30-second period from a distance of their own choosing, in close proximity to the basket. Each successful shot was awarded a value of one point. To assess the participants' passing abilities, they were instructed to execute a one-handed baseball pass from a distance of 12 metres to rectangles delineated on a wall. The rectangles were arranged in an overlapping configuration, with the smallest width of 50 cm, length of 25 cm, the central rectangle measuring 1 m by 60 cm, and the largest rectangle measuring 1.5 m by 1 m. A successful pass that struck the centre rectangle was awarded three points, two points for a pass that hit the middle rectangle, and one point for a pass that struck the outer rectangle. In order to assess the participants' ability to dribble, four obstacles were positioned at 180-cm intervals along a line. The distance between the initial obstacle and the starting line was 360 centimetres. Participants commenced the dribbling task from the starting line, navigating the obstacles and returning to the starting line within a specified time limit of 30 seconds. The total number of obstacles successfully negotiated was recorded as the score. The Johnson basketball skill test yielded four parameters: passing, shooting, dribbling, and the total score of the test.

AAHPERD basketball speed shooting test The participants commenced shooting at the starting line within the designated shot-testing area. The participants propelled their shots towards the hoop from the initial zone, allowing them to rebound the ball and subsequently dribble to the alternative shooting zone, where they proceeded to shoot. Each participant was required to shoot at least once from each of the five designated shooting zones, with at least one foot within the shooting zone at the time of shooting. Following unsuccessful attempts at shooting, participants were permitted to attempt a layup after the rebound. However, it was not permitted to attempt two consecutive layups. A maximum of four layups was permitted throughout the course of the test. The participant was required to execute a legal shot or layup from the five-shot zone until the "stop" signal was given. Upon the expiration of the 60-second interval, the speed shooting test was concluded. Successful shots and layups were recorded by the practitioner as two points. In the event of a failed shot that subsequently returned from the hoop, the participant was awarded one point. If a layup shot was successfully made after the ball had been controlled and subsequently rebounded, two points were awarded. In the event of two consecutive successful layup shots, no points were awarded for the second shot. A maximum of four layups could be attempted within the 60-second period. No points were awarded for layup shots attempted after the fourth shot. No points were awarded for shots that constituted rule violations, such as steps, ball carrying, and shooting line violations.

Statistical analyses At the end of the research, the Statistical Package for the Social Sciences (SPSS) software package was used for the statistical analysis of the obtained data. The data were presented as mean and standard deviation. The Shapiro-Wilk test was applied for normality, and the Levene test was used for homogeneity. Skewness and kurtosis values were checked for data sets that did not show a normal distribution, and data sets within ±2 were considered to have a normal distribution. The Mauchly sphericity test was used to test the sphericity assumption. The Greenhouse-Geisser correction was applied in measurements where the sphericity assumption was not met. A one-way analysis of variance (ANOVA) for repeated measures with a 95% confidence interval was applied to analyze the differences among the protocols. The least significant difference correction was used to determine in which specific protocols the differences occurred. Effect sizes were calculated using partial eta squared (ηp²) to determine the magnitude of observed differences. Statistical results were evaluated at a significance level of p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Basketball players had to be free of both chronic and acute upper respiratory tract infections, as well as any chest diseases.
* Participants had to have no history of smoking or other habits that could impair respiratory function.
* Participants had to provide written informed consent prior to the study.

Exclusion Criteria:

* Participants with any history of cardiovascular, pulmonary, or neuromuscular disorders that could affect respiratory function.
* Individuals who had undergone respiratory muscle training within the past six months.
* Athletes with any current musculoskeletal injury that could interfere with performance tests.
* Those who reported the use of medication affecting respiratory or neuromuscular function.
* Participants who were unable to complete all testing sessions due to personal reasons or external factors.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 10 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-06-10 (Actual); Study Completion 2023-06-11 (Actual)

PRIMARY OUTCOMES:
Johnson Basketball Skill Test | Measured immediately after each intervention session.
  Shooting ability was assessed by recording the number of successful shots made within 30 seconds from a self-selected position near the basket (1 point per shot). Passing ability was evaluated using a one-handed baseball pass from 12 meters toward a target wall with three overlapping rectangles (smallest: 50×25 cm, middle: 1×0.6 m, largest: 1.5×1 m). Passes scored 3, 2, or 1 point based on accuracy. Dribbling ability was measured using four obstacles spaced 180 cm apart, with participants weaving through and returning to the start within 30 seconds. The score was based on the number of obstacles successfully navigated. The Johnson Basketball Skill Test provided passing, shooting, dribbling, and total skill scores.
AAHPERD Basketball Speed Shooting Test | Measured immediately after each intervention session.
  Participants began shooting from the designated starting zone, moving between five shooting zones while maintaining at least one foot within the zone. Missed shots allowed a layup attempt after rebounding, but consecutive layups were restricted (max: 4 per test). The test lasted 60 seconds, and points were awarded as follows: 2 points for successful shots or layups, 1 point for missed shots rebounding off the hoop, and no points for rule violations (e.g., traveling, carrying, line violations). The test concluded upon the "stop" signal.

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziantep University, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: Unending
Access Criteria: The datasets generated and/or analysed during the current study are available in the Figshare repository.
URL: https://www.doi.org/10.6084/m9.figshare.28536197

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-01): https://cdn.clinicaltrials.gov/large-docs/16/NCT06894316/Prot_SAP_000.pdf